CLINICAL TRIAL: NCT03508804
Title: Lidocaine-Prilocaine Cream in Conjunction With Lidocaine Paracervical Block for Pain With First-Trimester Abortion: A Double-Blind Randomized Controlled Trial
Brief Title: Lidocaine-Prilocaine Cream in Conjunction With Paracervical Block for Pain With Abortion
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-38207
Record Dates: First submitted 2016-06-15; First posted 2018-04-26 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Pain
Keywords: surgical abortion; cervical anesthesia; pain control
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine-prilocaine cream (Experimental): 5-10 minutes prior to the start of the procedure, the participant will self-administer 10ml of the lidocaine-prilocaine cream vaginally using a syringe
  Interventions: Drug: Lidocaine-Prilocaine Cream; Drug: 1% Lidocaine Paracervical Block
- Placebo cream (pain lucubrating gel) (Placebo Comparator): 5-10 minutes prior to the start of the procedure, the participant will self-administer 10ml of the placebo cream vaginally using a syringe
  Interventions: Drug: Placebo Cream; Drug: 1% Lidocaine Paracervical Block

INTERVENTIONS:
Drug: Lidocaine-Prilocaine Cream — 10ml of vaginally self-administered cream composed of an eutectic mixture of 2.5% lidocaine, 2.5% prilocaine
  Other Names: EMLA
  Arms: Lidocaine-prilocaine cream
Drug: Placebo Cream — 10ml of vaginally self-administered placebo cream
  Arms: Placebo cream (pain lucubrating gel)
Drug: 1% Lidocaine Paracervical Block — Paracervical block of 10ml of 1% lidocaine

SUMMARY:
The investigators theorize that the application of a lidocaine-prilocaine cream 5-10 minutes prior to the administration of a paracervical block could decrease pain associated with its administration and pain with abortion overall.

DETAILED DESCRIPTION:
This is a superiority, double-blind randomized controlled trail of women ages 18 and older presenting for first-trimester surgical abortion. The lidocaine-prilocaine cream will be used in the experimental group in conjunction with a paracervical block, whereas plain lubricating gel will be used in conjunction with a paracervical block for the placebo, control group.

ELIGIBILITY:
Inclusion Criteria:

* surgical abortion patient at 5 0/7 to 11 6/7 weeks gestational age;
* English or Spanish speaking;
* ability to give informed consent

Exclusion Criteria:

* pre-operative use of misoprostol;
* allergy to study medications (lidocaine, prilocaine, versed, fentanyl);
* known uterine anomaly;
* prior cervical surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pain perceived as measured by a Visual Analog Scale (0-100mm) at the time of cervical dilation | Intraoperative; Immediately following cervical dilation

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No